CLINICAL TRIAL: NCT05195411
Title: Nephroblastoma With Vena Cava Thrombosis : Multicenter Study Over 20 Years - Analysis of Key Elements of Surgical Management
Brief Title: Vascular Thrombus Involvement in Nephroblastoma
Acronym: VIN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201331
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2023-11

CONDITIONS: Nephroblastoma With Vena Cava Thrombosis
Keywords: Nephroblastoma; Wilms tumor; Vena cava thrombosis; Surgical management
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nephroblastoma with vena cava thrombosis: Children with nephroblastoma with vena cava thrombosis +/- atrial extension, cared between 1999 and 2019 in Parisian hospitals: Necker and Bicêtre.

SUMMARY:
Nephroblastoma (Wilms tumor) is the most common kidney tumor in children. It is a malignant embryonic tumor with a good prognosis with more than 85% long-term survival with appropriate chemotherapy, surgery (which most often consists of a total nephrectomy) and radiotherapy for locally invasive forms. Some nephroblastomas (approximately 10%) present with vascular extension with vena cava thrombus, a situation which may worsen the prognosis due to the complexity of the surgery. While the oncological treatment of nephroblastoma is highly formalized, to date there is no specific guideline on the surgical management of this rare clinical presentation of nephroblastomas.

The aim of the study is to provide recommendations for the surgical management of nephroblastomas with vena cava thrombus in a large multicenter series.

DETAILED DESCRIPTION:
Nephroblastoma (Wilms tumor) is the most common kidney tumor in children. It is a malignant embryonic tumor with a good prognosis with more than 85% long-term survival with appropriate chemotherapy, surgery (which most often consists of a total nephrectomy) and radiotherapy for locally invasive forms. Some nephroblastomas (approximately 10%) present with vascular extension with vena cava thrombus, a situation which may worsen the prognosis due to the complexity of the surgery. While the oncological treatment of nephroblastoma is highly formalized, to date there is no specific guideline on the surgical management of this rare clinical presentation of nephroblastomas.

The management of children with nephroblastomas with vena cava thrombosis is very specific because of the vital risks to diagnosis, especially pulmonary embolism but also cardiac arrest (in the event of extension in the right atrium) and Cerebrovascular accidents by embolism, rarer. Surgery of the primary tumor and its intravascular extension is complex and may require the use of extracorporeal circulation, a source of significant morbidity and even mortality. These patients who will actually have a single kidney are at high risk for renal failure due to possible contralateral kidney damage during surgery. Surgery is not clearly codified because cases are rare, including in expert centers.

The aim of the study is to provide recommendations for the surgical management of nephroblastomas with vena cava thrombus in a large multicenter series.

ELIGIBILITY:
Inclusion Criteria:

* Minors with nephroblastoma with vena cava thrombosis +/- atrial extension.
* Cared between 1999 and 2019 in the centers of the study.

Exclusion Criteria:

- Other renal and non-renal tumors with vena cava thrombosis.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with nephroblastoma with vena cava thrombosis +/- atrial extension cared between 1999 and 2019 in Parisian hospitals: Necker and Bicêtre.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Survival | 22 years
  Study of the medical file.
Recurrence | 22 years
  Study of the medical file. Local or metastatic recurrence.
Determination of surgical management recommendations | 2 months
  Study of the medical file. Determination of surgical management recommendations based on survival, the occurrence of local or metastatic recurrence and the study of medical care of the patient.

SECONDARY OUTCOMES:
Intraoperative complications | 1 day
  Study of the medical file. Description of intraoperative complications and Dindo-Clavien classification (classification that defines and grades operative complications in 10 grades).
Post-operative complications | 30 days
  Study of the medical file. Description of post-operative complications and Dindo-Clavien classification (classification that defines and grades operative complications in 10 grades).
Long-term sequelae | 20 years
  Study of the medical file. Sequelae linked to the toxicity of chemotherapy, radiotherapy and surgery.
Identify the oncological and / or surgical prognostic risk factors | 2 months
  Study of the medical file. Identify the oncological and / or surgical prognostic risk factors depending on the medical treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Sarnacki, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Luca Pio, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pio L, Abib S, Guerin F, Chardot C, Blanc T, Sarrai N, Martelli H, De Souza FKM, Fanelli MCA, Tamisier D, Guilhen JCS, Le Bret E, Belli E, Fadel E, Cypriano MDS, Minard V, Pasqualini C, Schleiermacher G, Lemelle L, Rod J, Irtan S, Pistorio A, Gauthier F, Branchereau S, Sarnacki S. Surgical Management of Wilms Tumors with Intravenous Extension: A Multicenter Analysis of Clinical Management with Technical Insights. Ann Surg Oncol. 2024 Jul;31(7):4713-4723. doi: 10.1245/s10434-024-15232-w. Epub 2024 Apr 5. PMID 38578552